CLINICAL TRIAL: NCT00781131
Title: A Randomized, Placebo Controlled Trial of Pregabalin for Post-operative Pain in Women Undergoing Abdominal Hysterectomy
Brief Title: Trial of Pregabalin for Post-operative Pain in Women Undergoing Abdominal Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWK-4101-2007
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): Pregabalin 75 mg
  Interventions: Drug: Pregabalin
- 3 (Experimental): Pregabalin 150 mg
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — pregabalin 75 or 150 mg
  Arms: 2; 3
Drug: Placebo — lactulose placebo
  Arms: 1

SUMMARY:
We hypothesize that pregabalin will decrease post-operative pain scores and opioid use following abdominal hysterectomy compared to placebo. This study has been designed to determine if after an abdominal hysterectomy, the addition of pregabalin to their peri-operative analgesia regimen will demonstrate superior analgesia compared to placebo in terms of lower pain scores and reduced usage of opioids. The primary outcome will be post-operative pain, measured by total opioid consumption.

Do women undergoing an abdominal hysterectomy with general anesthesia and receiving pregabalin prior to their surgery and 12 hours later have lower opioid consumption in the first 24 hours after their surgery than those women who received placebo?

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesia physical status class I & II
2. Age > 18 years
3. English-speaking
4. Capability to operate a patient-controlled analgesia (PCA) device

Exclusion Criteria:

1. Known or suspected allergy, sensitivity, or contraindication to pregabalin or any of the standardized medications (i.e. morphine, anesthetic agents)
2. Morbid Obesity (Body Mass Index ≥ 45 kg/m2)
3. History of a seizure disorder
4. Current therapy with pregabalin, gabapentin, or any opioid
5. Any other physical or psychiatric condition which may impair their ability to cooperate with post-operative study data collection
6. CrCl < 60 ml/min [CrCl = 0.85 x ((140 - age) x weight(kg)) / (72 x Cr(mg/dL)))]

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Do women undergoing an abdominal hysterectomy with general anesthesia and receiving pregabalin prior to their surgery and 12 hours later have lower opioid consumption in the first 24 hours after their surgery than those women who received placebo? | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] George RB, McKeen DM, Andreou P, Habib AS. A randomized placebo-controlled trial of two doses of pregabalin for postoperative analgesia in patients undergoing abdominal hysterectomy. Can J Anaesth. 2014 Jun;61(6):551-7. doi: 10.1007/s12630-014-0147-4. Epub 2014 Mar 26. PMID 24668315